CLINICAL TRIAL: NCT03505944
Title: Venetoclax, Lenalidomide and Rituximab in Patients With Relapsed/Refractory Mantle Cell Lymphoma
Acronym: VALERIA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-MCL7; 2017-001060-38 (EudraCT Number)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Relapsed Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Venetoclax+lenalidomide+rituximab
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — venetoclax + lenalidomide + rituximab

SUMMARY:
Phase I/II trial, with the aim of evaluating the efficacy of venetoclax to the backbone of rituximab-lenalidomide in patients with relapsed/refractory MCL.

ELIGIBILITY:
Inclusion criteria

* Age >18 years
* Histologically confirmed (according to the WHO 2016 classification) mantle cell lymphoma stage I-IV

  * Who have received at least 1 prior rituximab-containing chemotherapy regimen, with documented relapse or disease progression following the last anti-MCL treatment OR
  * Are not considered to be candidates for chemotherapy due to frailty or comorbidity
* At least 1 measurable site of disease (>1.5 cm long axis)
* WHO performance status 0 - 3
* Written informed consent.
* Female subjects of childbearing potential must (see page 52 for definition of not fertile):

  * Understand that the study medication is expected to be teratogenic
  * Agree to use, and be able to comply with, highly effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea.
  * All fertile women must agree to perform monthly pregnancy tests while on study medication and until 4 weeks after completion of study drug. Tests must have a minimum sensitivity of 25 mIE/ml and be medically witnessed
  * Highly effective contraception include:

Implant* Levonorgestrel-releasing intrauterine system (IUS)* Medroxyprogesterone acetate depot Tubal sterilisation Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses Ovulation inhibitory progesterone-only pills (i.e., desogestrel) NB! Patients using a hormonal method, must also use a second barrier method. Sexual abstinence (if refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the preferred and usual lifestyle of the subject).

* Male subjects must

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* All subjects must

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator

Exclusion criteria

* Chemotherapy or radiotherapy within 3 weeks
* Therapeutic antibodies or BTK inhibitors within 4 weeks
* Radioimmunotherapy within 10 weeks
* Major surgery within 4 weeks of inclusion in this trial.
* Previous treatment with venetoclax
* Impaired liver function: AST and ALT >3.0 × the upper normal limit (ULN) of institution's normal range; Bilirubin > 1.5 × ULN. Subjects with Gilbert's Syndrome may have a bilirubin > 1.5 × ULN, per discussion between the investigator and medical monitor. Elevated Bilirubin due to haemolytic anemia or caused by lymphoma, is not an exclusion criterion.
* Absolute neutrophil count (ANC) <1.0x 109, unless caused by bone marrow infiltration by lymphoma.
* Platelet count <60 x 109, unless caused by bone marrow infiltration by lymphoma.
* Creatinine clearance below 50 ml/min (Cockcroft-Gault)
* Known CNS lymphoma.
* Heart failure in NYHA stage IV or other serious CVD
* Pulmonary failure (ex chronic disease with hypoxemia)
* Active serious infections such as hepatitis B or C and HIV
* Conditions with serious immunocompromised state
* Breastfeeding women must be excluded or stop breastfeeding
* Other active malignancy.
* Psychiatric illness or condition which could interfere with the subjects' ability to understand the requirements of the study.
* Requirement of corticosteroid therapy at a dose >10 mg prednisolone/day.
* Hypersensitivity to venetoclax, lenalidomide or rituximab, or HACA against rituximab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  The primary objective is to assess the overall response rate (ORR) at 6 months with lenalidomide-venetoclax and rituximab, in patients with relapsed or refractory mantle cell lymphoma, by use of an MRD driven strategy. ORR includes complete (CR) and partial remissions (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, Principal Investigator — Skane University Hospital
Locations (17):
- Denmark (5):
  - Department of Hematology Aalborg University Hospital, Aalborg
  - Department of Hematology Aarhus University Hospital, Aarhus
  - Clinic of Hematology L-4241 Rigshospitalet, Copenhagen
  - Department of Hematology X Odense University Hospital, Odense
  - Hæmatologisk Afdeling Zeeland University Hospital, Roskilde, Roskilde
- Finland (3):
  - Department of Hematology Helsinki University Hospital Comprehensive Cancer Center, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Norway (3):
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - St. Olav Hospital, Trondheim
- Sweden (6):
  - Department of Hematology Linköping University Hospital, Linköping
  - Department of Medicine Sunderbyn Hospital, Luleå
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Department of Oncology Norrland University Hospital, Umeå
  - Uppsla Academic Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jerkeman M, Kolstad A, Hutchings M, Pasanen A, Meriranta L, Niemann CU, Kragh Jorgensen RR, El-Galaly TC, Riise J, Leppa S, Christensen JH, Sonnevi K, Pedersen LB, Wader KF, Glimelius I. MRD-driven treatment with venetoclax-R2 in mantle cell lymphoma: the Nordic Lymphoma Group MCL7 VALERIA trial. Blood Adv. 2024 Jan 23;8(2):407-415. doi: 10.1182/bloodadvances.2023011920. PMID 38113470